CLINICAL TRIAL: NCT06995664
Title: Partial Volume High-Dose Irradiation in Renal Cell Carcinoma for Intra-TUmoural Control ALongside Current Management - a Randomised Feasibility Study
Brief Title: Partial Volume High-Dose Irradiation in Renal Cell Carcinoma for Intra-TUmoural Control ALongside Current Management
Acronym: VIRTUAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5652
Record Dates: First submitted 2024-08-12; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma; Renal Cell Carcinoma Metastatic
Keywords: standard palliative dose radiotherapy; high-dose hypofractionated radiotherapy; radiotherapy; unblinded
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: 2 treatment arms, patients randomised 1:1; no cross-over
Masking Description: Unblinded to investigator and participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard palliative-dose radiotherapy, 30Gy in 10 fractions in 3Gy per fraction over 2 weeks
- Experimental / High-dose (Experimental): High-dose radiotherapy, 30Gy in 5 fractions in 6Gy per fraction on alternate days/2-3 fractions a week over 2 weeks
  Interventions: Procedure: radiotherapy

INTERVENTIONS:
Procedure: radiotherapy — External Beam Radiotherapy - hypofractionated, short radiotherapy regime of 30Gy in 5 fractions (6Gy per fraction) delivered on alternate days over 2 weeks
  Arms: Experimental / High-dose

SUMMARY:
Prospective, randomised, feasibility study of patients with localised or metastatic renal cell carcinoma (RCC) comparing standard palliative dose radiotherapy to a high-dose hypofractionated regime.

Primary aim

• To demonstrate feasibility of a randomised study comparing high-dose hypofractionated radiotherapy versus standard palliative dose radiotherapy in localised or metastatic renal cell carcinoma The aim is to recruit a minimum of 24 patients; 12 to the control arm and 12 to the high-dose regime.

2 treatment arms, no placebo:

* Control arm - standard palliative-dose radiotherapy, 30Gy in 10 fractions in 3Gy per fraction over 2 weeks
* High-dose arm - high-dose radiotherapy, 30Gy in 5 fractions in 6Gy per fraction on alternate days/2-3 fractions a week over 2 weeks

DETAILED DESCRIPTION:
HYPOTHESIS The investigators hypothesise that it is feasible to recruit to a study of localised and metastatic renal cell carcinoma comparing a high-dose short fractionation radiotherapy regime (30Gy in 5 fractions in alternate day fractions over 2 weeks) in comparison to the standard palliative dose-fractionation (30Gy in 10 fractions in daily fractions over 2 weeks).

AIMS Primary aim

• To demonstrate feasibility of a randomised study comparing high-dose hypofractionated radiotherapy versus standard palliative dose radiotherapy in localised or metastatic renal cell carcinoma

Secondary aim

* To report acute and late toxicity in both treatment groups
* To demonstrate completion of quality of life (QOL) validated EORTC forms by patients under study

STUDY DESIGN

* Randomised 1:1
* The study is unblinded for the trial investigators and participants.

VISITS (in line with routine standard care):

* 1 Pre-treatment appointment
* 1 CT planning scan (immobilisation/mould room as required dependent on anatomical site)
* 10 radiotherapy treatment appointments (Control Arm) / 5 radiotherapy treatment appointments (Experimental Arm)
* 2 on-treat clinic reviews (week 1 and week 2)
* End of Treatment/Safety follow up (4 weeks post-radiotherapy)
* Follow-up at 3 months, 6 months, and 12 months

INVESTIGATIONS

* Quality of Life questionnaires
* Blood tests
* Clinical/Physical Examination

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma (RCC) (histological confirmation of metastasis not required) or clinically consistent with RCC as per multidisciplinary team (MDT) diagnosis.
* Not suitable for surgical resection, metastasectomy or ablative therapy due to tumour or patient factors
* All extracranial sites which clinically require radiotherapy (as per clinician discretion)
* Age ≥18 years
* Karnofsky Performance Status (KPS) ≥50
* Adequate baseline organ function applicable to site-of irradiation
* Haemaglobin ≥90g/dl
* Platelets ≥50
* Bilirubin <3x ULN
* INR <1.4 or correctable with vitamin K
* AST or ALT <5x normal range
* Creatinine <200umol/L (or established on dialysis). Note patients on dialysis are unable to have dynamic contrast enhanced MRI.
* The use of concurrent systemic therapy is acceptable
* Ability of the research subject to understand and the willingness to sign a written informed consent document
* Able to undergo all mandated staging and follow-up investigations
* Negative pregnancy test (for women of childbearing potential)

Exclusion Criteria:

* Expected prognosis <6 months
* Uncontrolled intracranial metastases
* Previous radiotherapy, such that the delivery of further radiotherapy is not feasible
* Unable to have necessary radiotherapy planning, radiotherapy related investigations/fiducials (if required)
* Co-morbidities or any psychological, familial, sociological or geographical condition which may preclude ability to undergo/attend investigations, treatment or follow-up
* Other active primary cancer
* Pregnant or lactating
* Requiring ongoing treatment with a concomitant medication, which is contraindicated alongside radiotherapy (e.g. methotrexate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 24 months
  To demonstrate feasibility of recruitment (assessed by 35% of eligible patients accepting the offer of recruitment). To calculate the proportion of patients that accept the offer of recruitment to the study. The denominator is the number of eligible patients that have been approached for the study

SECONDARY OUTCOMES:
Secondary aim | 24 months
  To evaluate acute ≥Grade 3 CTCAE v5.0 toxicity by treatment group. 'Acute' is defined as less than or equal to 3 months post-completion of radiotherapy.
Secondary aim | 24 months
  To evaluate late ≥Grade 3 CTCAE v5.0 toxicity by treatment group. 'Late' is defined as over 3 months from completion of radiotherapy.
Secondary aim | 24 months
  To demonstrate completion of quality of life (QOL) validated EORTC forms by patients under study, by reporting upon the proportion of patients completing quality of life (QOL) questionnaires at baseline and follow up

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHSFT, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No